CLINICAL TRIAL: NCT03685877
Title: Profile of Hypocalcemia in Infants and Children Admitted to Assiut University Children Hospital
Brief Title: Hypocalcemia in Infants and Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Fathy Farghali, Profile of hypocalcemia in infants and children admitted to Assiut University Children Hospital., Assiut University
Other Study IDs: HCIIC
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-09

CONDITIONS: Hypocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypocalcemia is defined as reduction in the level of the ionized calcium in the blood to less than 0.95 mmole/ litre.

In some cases it is associated with symptoms such as neuromuscular impairment in the form of convulsions ,carpopedal spasm,parathesia ,laryngiospasm ,stridor……etc .Calcium circulates in blood stream in three fractions :protein bound to calcium,primarly to albumen(40%) and in 50% of the cases calcium is present in the ionized state which is physiologically active (Dias ,c et a l, 2013) . Symptomatizing hypocalcemia may occur in cases of vitamin D deficiency rickets (nutritional deficiency in infants less than two years ) .It may also occur in vitamin D resistant rickets e.g renal rickets because of failure of the kidney to synthesize 1-OH cholecalciferol of the 1-25 di-OH cholecalciferol (the active form of vitamin D).

DETAILED DESCRIPTION:
Hypocalcemia is defined as reduction in the level of the ionized calcium in the blood to less than 0.95 mmole/ litre.

In some cases it is associated with symptoms such as neuromuscular impairment in the form of convulsions ,carpopedal spasm,parathesia ,laryngiospasm ,stridor……etc .Calcium circulates in blood stream in three fractions :protein bound to calcium,primarly to albumen(40%) and in 50% of the cases calcium is present in the ionized state which is physiologically active (Dias ,c et a l, 2013) . Symptomatizing hypocalcemia may occur in cases of vitamin D deficiency rickets (nutritional deficiency in infants less than two years ) .It may also occur in vitamin D resistant rickets e.g renal rickets because of failure of the kidney to synthesize 1-OH cholecalciferol of the 1-25 di-OH cholecalciferol (the active form of vitamin D). In some cases the liver fails to synthesize the 25-OH group of the active 1-25 di hydroxy cholecalciferol . In cases of malabsorption hypocalcemia may occur because of lack of absorption of both calcium and vitamin D from the gastrointestinal tract.

Symptomatizing Ionized hypocalcemia has been reported as an early event associated with organ dysfunction in children admitted to intensive care unit. This suggests that hypocalcemia may occur in association with other causes than those mentioned above. It has been reported in cases with sepsis, shock and in association with the use of anticonvulsants. It may occur in cardiac arrythmia and tetany (Khadilkar,V & Khadilkar,V,2017).

Regulation of calcium haemostasis is done by two principle hormones: vitamin D and parathyroid hormone.

These hormones act on three target organs: the intestine, the kidney and bones. In cases of advanced vitamin D deficiency rickets and in cases of vitamin D resistant rickets compensatory hyperparathyroidism may occur.( Basatemur & Sutcliffe,2015) Research question: to find out the causes and differential diagnosis of syptomatizing hypocalcemia in infants and children admitted to Assiut University Children Hospital using the available datafrom the literature.

The current strategy for dealing with this problem will be described using an algorithm covering the various clinical presentations and investigations to reach the final diagnosis guided by( Fukomoto,S et al,2008 , Pacaud,D & Dawrant ,J,2007 as well as Kelly,A & Levine,M,2013)

ELIGIBILITY:
Inclusion Criteria:

* All symptomatizing hypocalcemic cases presenting acutely to the Assiut University Children Hospital with convulsions, carpopedal spasm, stridor, renal symptoms or malabsorption symptoms aged > 1 month to the age of 17 years.

Exclusion Criteria:

* All neonatal hypocalcemic cases.

Ages: 1 Month to 17 Years | Sex: All
Age Groups: Child
Study Population: : All data will be collected in a sheet form for all cases of acutely symptomatizing hypocalcemia admitted during period from 1st November 2018 to End of November 2019.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-30 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
hypocalcemia in infants and children | 1YEAR
  Good management of all cases with symptomatizing hypocalcemia admitted at Assiut University Children Hospital based on knowing the exact final diagnosis by knowing the result of the various investigations as indicated

SECONDARY OUTCOMES:
pediatric hypocalcemia | 1YEAR
  Recommendation for Assiut University Children Hospital for providing all the investigation required so that the patient will not need to pay for any of them if they are not done in the inpatient of the pediatric Assiut University Children Hospital at the present time of the research.

IPD SHARING:
Plan to Share IPD: Undecided